CLINICAL TRIAL: NCT06609863
Title: dTACE-HAIC Combined With Bevacizumab and Atezolizumab for Huge Intermediate and Advanced Hepatocellular Carcinoma: a Prospective Phase II Study
Brief Title: dTACE-HAIC Combined With Bevacizumab and Atezolizumab for Huge Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Liver Projiect 9
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Advanced Hepatocellular Carcinoma; Atezolizumab; Bevacizumab; Chemotherapy
Keywords: hepatocellular carcinoma; Atezolizumab; Bevacizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dTACE-HAIC plus Bevacizumab and Atezolizumab (Experimental): dTACE procedure was a 2.8-F microcatheter was super-selectively inserted into the tumor feeding artery using the coaxial technique. Then drug-eluting microspheres was used (100-300um, 300-500um). Hepatic arterial infusion of oxaliplatin, fluorouracil, and leucovorin every 4 weeks. Lenvatinib 12 mg (or 8 mg) once daily (QD) oral dosing. Toripalimab, 200 mg intravenously every 2 weeks.
  Interventions: Procedure: dTACE-HAIC

INTERVENTIONS:
Procedure: dTACE-HAIC — dTACE procedure was a 2.8-F microcatheter was super-selectively inserted into the tumor feeding artery using the coaxial technique. Then drug-eluting microspheres were used (100-300um). The microcatheter was reserved at the proper/left/right hepatic artery according tumor location. After the patient returned to the ward, the following FOLFOX-based regime was intra-arterially administered through the microcatheter. The FOLFOX regimen was administered via the hepatic artery as follows: 85 or 135 mg/m2 oxaliplatin from hour 0 to 2 on day 1, and 400 mg/m2 leucovorin from hour 2 to 4 on day 1, and 400 mg/m2 fluorouracil bolus at hour 5 on the day 1; and 2400 mg/m2 fluorouracil over 46 h on days 1 and 2. Hepatic arterial infusion chemotherapy administration of oxaliplatin, fluorouracil, and leucovorin via the tumor feeding arteries every 4 weeks

SUMMARY:
This study intends to evaluate the efficacy and safety of drug-eluting transcatheter arterial embolization-hepatic arterial infusion chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin (dTACE-HAIC) plus Bevacizumab and Atezolizumab for patients with intermediate-advanced huge hepatocellular carcinoma.

DETAILED DESCRIPTION:
Drug-eluting transcatheter arterial embolization (dTACE) and hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin, 5-fluorouracil and leucovorin are effective and safe for hepatocellular carcinoma. Atezolizumab + Bevacizumab was superior to sorafenib in overall survival in advanced hepatocellular carcinoma. The anti-VEGF combined programmed cell death protein-1 legend 1 (PD-L1) inhibitor were effective and tolerable in patients with advanced hepatocellular carcinoma. We aimed to describe the efficacy and safety of locoregional therapy (dTACE/HAIC) combined with Bevacizumab and Atezolizumab inhibitor in patients with huge hepatocellular carcinoma who can not receive radical therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of HCC.
2. Age between 18 and 75 years;
3. The maximum tumor size ≥10 cm;
4. Intermediate-advanced huge HCC, advanced HCC with PVTT type I-III
5. limited metastases (≤5).
6. Child-Pugh class A or B;
7. Eastern Cooperative Group performance status (ECOG) score of 0-1;
8. Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 32 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3
9. Prothrombin time ≤18s or international normalized ratio < 1.7.
10. Ability to understand the protocol and to agree to and sign a written informed consent document.

Exclusion Criteria:

1. Diffuse HCC;
2. Extrahepatic metastasis >5;
3. Obstructive PVTT involving mesenteric vena cava (PVTT IV).
4. Serious medical comorbidities.
5. Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
6. untreated or incompletely treated esophageal or gastric varices (assessed with esophagogastroduodenoscopy) with bleeding or high risk of bleeding.
7. Eastern Cooperative Group performance status (ECOG) score of ≥2;
8. Known or suspected allergy to the investigational agents or any agent given in association with this trial.
9. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
10. Evidence of bleeding diathesis.
11. Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all included patients whose best overall response (BOR) is either a complete response or partial response.

SECONDARY OUTCOMES:
Progression-Free-Survival (PFS) | 12 months
  PFS is the length of time from the date of inclusion until tumor progression.
Overall survival (OS) | 24 months
  OS is the length of time from the date of inclusion until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Duan, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General hospital, Beijing, None Selected, China